CLINICAL TRIAL: NCT01351272
Title: Genetic Modulation of Functional Brain Activity of Attention-deficit/Hyperactivity Disorder-related Working Memory Processes
Brief Title: Genetic Modulation of Working Memory in Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: BEAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Martin Herrmann, Principal Investigator, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: W004PS0108_1
Record Dates: First submitted 2011-04-29; First posted 2011-05-10 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylphenidate, non-retard (Experimental)
  Interventions: Drug: Methylphenidate, non-retard
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate, non-retard — Medication (methylphenidate, non-retard) will be titrated to optimal response within 6 weeks, with a maximum of 10 mg/day in week 1, 20 mg/day in week 2, 30 mg/day in week 3, 40 mg/day in week 4, 50 mg/day in week 5, and 60 mg/day in week 6, unless adverse effects emerged. After successful adjustment, medication will be maintained until week 6. Dosing will be based on at least two-weekly evaluations by a psychiatrist, including an interview with a review of symptoms and side effects, completion of the Clinical Global Impression (CGI) scale and completion of a standardised Side Effects Rating Scale for psychostimulants (SERS). The maximal daily dosage of MPH is 60 mg. Within this double blind study the same procedure is applied for the placebo condition.
  Arms: methylphenidate, non-retard
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study the investigators will measure the functional brain activity of adult Attention Deficit Hyperactivity Disorder (ADHD) patients, genotyped according to the COMT genotype, during a Working Memory Paradigm, before and after a placebo controlled treatment with MPH for 6 WEEKS. Within this design, the investigators will be able to evaluate the therapeutic effect of MPH treatment on cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Only participants will be included who (1) fulfil the diagnostic criteria defined in guidelines for the diagnosis of ADHD in childhood and adulthood and who (2) would be treated with MPH also for clinical indications outside the study.
* Provision of written informed consent
* A diagnosis of a ADHD (314.xx) by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
* Females and males aged 18-50 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
* Able to understand and comply with the requirements of the study
* Right-handed according Edinburgh Handedness Inventory (Oldfield, 1971)
* German as first language
* Caucasian ethnicity

Exclusion Criteria:

* Pregnancy or lactation; women capable of childbearing are required to use a reliable method (Pearl-index < 1%) of contraception (e.g. hormonal treatment, intrauterine device, vasoligation in the partner, sexual abstinent)
* Any current DSM-IV Axis I disorder not defined in the inclusion criteria requiring current additional treatment
* Motoric tics, siblings with tics or positive family history or diagnosis of a Tourette syndrome
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to methylphenidate, as judged by the investigator
* Present pre-treatment with methylphenidate (within the last three month prior to study treatment)
* Intake of MAO-inhibitors within the last 14 days prior to study treatment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. Congestive Heart Failure / CHF, angina pectoris, hypertension, narrow angle glaucoma, hyperthyroidism, thyreotoxicosis, cardiac arrhythmia, cardiac infarction) as judged by the investigator.
* Epilepsy
* An absolute neutrophil count (ANC) of minor 1.5 x 10 exp 9 per litre
* Involvement in the planning and conduct of the study
* Previous enrolment or randomisation of treatment in the present study
* Participation in another drug trial within 4 weeks prior to enrolment into this study
* Moderate, severe, or profound mental retardation
* Heart pacemakers, cochlea implants, other metal parts in the head outside the mouth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Psychiatrie, Psychosomatics and Psychotherapy, Würzburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start: May 2011 Primary Completion: December 2012 Study Completion: March 2013 Wuerzburg University Hospital
Groups:
- Control: Placebo: For placebo treatment the same procedure was applied like in the verum condition
Period: Overall Study
Arm/Group | Methylphenidate, Non-retard | Control: Placebo
Started | 19 | 16
Completed | 14 | 13
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate, Non-retard | Control: Placebo | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (9.7) | 35.3 (10.2) | 36.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation
Description: Functional brain activity in right Superior Frontal Gyrus (SFG) during the working memory task post treatment as measured by fMRI. For each participant and conditions the estimated parameters are metric, and can be further analysed with ANOVAs or t-tests.
Time Frame: 6 weeks
Population: lost of data due to fmri specific issues
Measure: Mean (Standard Error); unit: Beta weights of contrast
Arm/Group | Methylphenidate, Non-retard | Control: Placebo
Number analyzed (Participants) | 14 | 13
Beta weights of contrast | 0.19 (0.09) | -0.08 (0.08)
Statistical Analysis 1: Comparison: Methylphenidate, Non-retard vs Control: Placebo; Test type: Superiority; p = 0.09, SPM two-sample t-test

2. Secondary Outcome: Neuropsychology
Description: Accuracy for the working memory paradigm at post. Accuracy was defined as the ratio of correct responses (correctly pressed and correctly not pressed) to total number of stimuli. Higher values indicate better perfromance.The theoretical range goes from 0 to 1.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: accuracy index
Arm/Group | Methylphenidate, Non-retard | Control: Placebo
Number analyzed (Participants) | 10 | 11
accuracy index | 0.97 (0.03) | 0.98 (0.01)
Statistical Analysis 1: Comparison: Methylphenidate, Non-retard vs Control: Placebo; Test type: Superiority; p = 0.16, t-test, 1 sided

3. Secondary Outcome: ADHD Core Symptoms: Measured by Conners Adult ADHD Rating Scales (CAARS), Inattention Scale
Description: Changes in CAARS scale ( T-values, 50 indicates the population mean with a standard deviation of 10) from pre to post.
  Higher T values indicate higher symptoms. T-score over 60 indicates clinically relevant ADHS symptoms
  More negative values of the difference indicate higher symptom reduction, therefore a better outcome.
  Range of T-values for pre and post measurements between 35 and 90, potential range for differences -55 to +55
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Methylphenidate, Non-retard | Control: Placebo
Number analyzed (Participants) | 19 | 15
T-score | -18.9 (3.76) | -12 (4.44)
Statistical Analysis 1: Comparison: Methylphenidate, Non-retard vs Control: Placebo; Test type: Superiority; p = 0.09, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: through study completion at day 70
Arm/Group | Methylphenidate, Non-retard | Control: Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/16
Other Adverse Events (participants affected / at risk) | 18/19 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate, Non-retard (N=19) | Control: Placebo (N=16)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate, Non-retard (N=19) | Control: Placebo (N=16)
Headache (Nervous system disorders) | 10 (12) | 4 (4)
Therapeutic apical closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Labile blood pressure (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pain in throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness postural (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Feeling agitated (Psychiatric disorders) | 1 (1) | 0 (0)
Difficulty sleeping (Psychiatric disorders) | 1 (3) | 2 (2)
Infection of gastrointestinal tract (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 1 (1)
menstrual problem (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (4)
cramp (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
low back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rupture of meniscus of knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
common cold (Infections and infestations) | 6 (8) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes